CLINICAL TRIAL: NCT02330081
Title: Mirasol System for Whole Blood: Survival and Recovery of Radio-labeled Platelets Derived From Mirasol-treated Whole Blood in Healthy Volunteers
Brief Title: Survival and Recovery of Radio-labeled Platelets Derived From Mirasol-treated Whole Blood
Acronym: Medic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo BCTbio (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CTS-0081
Record Dates: First submitted 2014-12-30; First posted 2015-01-01 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Blood Safety
Keywords: pathogen reduction technology; whole blood; Platelets; Mirasol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mirasol (Experimental): Subject will be infused with two products at the same time:
  1. radio-labeled platelets derived from subjects stored whole blood which has been treated with Mirasol.
  2. radio-labeled platelets derived from subjects untreated fresh whole blood.
  Interventions: Device: Mirasol treatment of whole blood

INTERVENTIONS:
Device: Mirasol treatment of whole blood — Subject will be infused with two products at the same time:
  1. radio-labeled platelets derived from subject's stored whole blood which has been treated with Mirasol.
  2. radio-labeled platelets derived from subject's untreated fresh whole blood.
  Other Names: Mirasol pathogen reduction system; Mirasol system for whole blood

SUMMARY:
A total of twelve healthy volunteers will donate one unit of fresh whole blood. This unit will be treated with the Mirasol Pathogen Reduction Technology for Whole blood and then stored for 24h. At the end of storage, platelet concentrates will be separated from the unit, tested for key in vitro parameters and radiolabeled. On the same day (so 24h after the donation of whole blood), the volunteer will donate a fresh sample of whole blood. Platelets will be separated from this fresh sample and labeled with another radio-isotope. Then, the two radiolabeled platelet aliquots will be infused simultaneously and the recovery and survival of the two types of platelets will be measured.

DETAILED DESCRIPTION:
The study will be a prospective, single-center, single-arm, intra-subject controlled, open-label design.

Subjects will donate one unit of fresh whole blood. This unit will be treated with the Mirasol PRT System for whole blood and then stored for 24 hours ± 1 hour at 22 ± 2°C. At the end of storage, platelet concentrates will be separated from the unit according to the Biomedical Excellence for Safer Transfusion (BEST) procedures. An aliquot will be removed from the platelet concentrates for testing and for radiolabeling and reinfusion. The platelets in Mirasol-treated whole blood will be tested for key in vitro parameters directly after treatment (Day 0) and at the end of storage (Day 1). Sterility testing will also be conducted on the stored units.

An aliquot of the platelet concentrate separated from each unit of stored Mirasol-treated whole blood will be radiolabeled with either 111Indium Oxine or 51Chromium, and autologously infused. An intra-subject control will be utilized as per the BEST guidelines for platelet radiolabeling procedures. On the day of infusion, the subject will donate a fresh sample of whole blood. Platelets will be separated from this fresh sample and labeled with the radio-isotope that was not used to label the subject's Mirasol-treated platelet sample. The two radiolabeled platelet aliquots (Mirasol-treated and fresh control) will be infused simultaneously, and the recovery and survival of the two types of platelets will be measured according to standard institutional practice.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult subjects, who meet the inclusion criteria defined by the Blood Center for whole blood donation.
2. Age ≥ 18 and < 70 years
3. Able to commit to the study follow-up schedule.
4. Subjects must have adequate antecubital venous access for whole blood collection and follow-up blood draws.
5. Subjects of child-bearing potential (female or male) must agree to use effective contraception per site guideline or abstain from heterosexual intercourse during the course of the study.
6. Female of childbearing potential must be willing to take a pregnancy test prior to infusion of radiolabeled platelets.
7. Subjects must agree to report adverse events (AEs) during the required reporting period.

Exclusion Criteria:

1. Use of medications that interfere with platelet function within 48 hours of planned whole blood collection.
2. Participation currently, or within the last 12 months, in another investigational trial that would potentially interfere with the analysis of this investigation (e.g., pharmaceutical).
3. Inability to comply with the protocol in the opinion of the investigator.
4. Unable or unwilling to give informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ray Goodrich, PhD, Study Chair — Terumo BCT VP Science, Clinical and Laboratory
Locations (1):
- Haukeland University Hospital, Bergen, Norway

RESULTS

PARTICIPANT FLOW:
Groups:
- Mirasol: Subject will be infused with two products at the same time:
  1. radio-labeled platelets derived from subjects stored whole blood which has been treated with Mirasol.
  2. radio-labeled platelets derived from subjects untreated fresh whole blood.
  Mirasol treatment of whole blood: Subject will be infused with two products at the same time:
  1. radio-labeled platelets derived from subject's stored whole blood which has been treated with Mirasol.
  2. radio-labeled platelets derived from subject's untreated fresh whole blood.
Period: Overall Study
Arm/Group | Mirasol
Started | 22
Completed | 14
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Donation did not meet criteria | 1
Not completed — Protocol Violation | 6

BASELINE CHARACTERISTICS:
Population: Modified Intent to Treat population (mITT) = all enrolled subjects who signed consent and have valid data (excluding Subjects V01 through V08 who had irreparably confounded data due to a calibration error of the radioactivity detection device). Additionally, subjects V01 and V08 exited the study prior to reinfusion of their radiolabeled platelets.
Arm/Group | Mirasol
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (11.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Norway | 14
Height [Mean (Standard Deviation); unit: cm] | 172.6 (9.08)
Weight [Mean (Standard Deviation); unit: kg] | 78.7 (13.68)
Blood type [Number; unit: participants]
  A | 6
  B | 1
  AB | 0
  O | 7
Rhesus status [Number; unit: participants]
  Positive | 14
  Negative | 0

OUTCOME MEASURES:

1. Primary Outcome: Platelet 24-hour Relative Recovery
Description: Relative recovery of platelets derived from Mirasol-treated whole blood (WB) units that had been stored for 24 ± 1 hours at 22 ± 2ºC, measured as a percentage of platelets derived from freshly collected WB from the same participant. Platelets were isolated from both Mirasol-treated WB and from fresh WB from the same participant, radiolabeled with either 111Indium or 51Chromium, and these 2 radiolabeled platelet samples (ie, 1 untreated, fresh and 1 Mirasol-treated, stored) were combined and reinfused back to the same participant.
Time Frame: 24 hours
Population: Per Protocol Population = all subjects in the mITT Population who met all of the inclusion and none of the exclusion criteria at enrollment, had no concurrent illness or notable signs/symptoms during the 24 hours prior to reinfusion, had completed all postinfusion blood sampling for recovery and survival calculations and had no protocol violations.
Measure: Mean (95% Confidence Interval); unit: Percentage of platelet count
Groups:
- Test Platelets From Mirasol-treated Whole Blood: Mirasol-treated platelets: Platelets were collected from 1 Test unit of whole blood that had been treated with the Mirasol pathogen reduction process and stored for 24 hours.
- Control Platelets: Control platelets: An aliquot of platelets derived from a freshly collected whole blood sample
Arm/Group | Test Platelets From Mirasol-treated Whole Blood | Control Platelets
Number analyzed (Participants) | 14 | 14
Percentage of platelet count | 43.31 [37.93 to 48.69] | 52.01 [45.22 to 58.80]
Statistical Analysis 1: Comparison: Test Platelets From Mirasol-treated Whole Blood vs Control Platelets; Test type: Non-Inferiority — The FDA validation level requirements for test platelet quality is that the lower 1-sided 95% confidence limit of platelet recovery must be ≥ 66% of fresh control platelet values; Risk Ratio (RR) = 83.3, 95% CI 1-sided [lower limit 76.2], Standard Error of Mean 4.97 — Estimate is the ratio of the mean platelet recovery of treatment over control

2. Primary Outcome: Relative Platelet Survival
Description: Mean survival time of platelets derived from Mirasol-treated whole blood (WB) units that had been stored for 24 ± 1 hours at 22 ± 2ºC as compared to the mean survival time of fresh platelets from the same donor, measured in hours. Platelets were isolated from both Mirasol-treated WB and from fresh WB from the same participant, radiolabeled with either 111Indium or 51Chromium, and these 2 radiolabeled platelet samples (ie, 1 untreated, fresh and 1 Mirasol-treated, stored) were combined and reinfused back to the same participant.
Time Frame: Days 1 through 10 post-infusion
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Test Platelets From Mirasol-treated Whole Blood | Control Platelets
Number analyzed (Participants) | 14 | 14
hours | 152.9 [136.4 to 169.4] | 188.8 [175.2 to 202.3]
Statistical Analysis 1: Comparison: Test Platelets From Mirasol-treated Whole Blood vs Control Platelets; Test type: Non-Inferiority — One of the FDA validation level requirements for test platelet quality is that the lower 1-sided 95% confidence limit of the mean platelet survival time must be ≥58% of fresh control platelet mean survival time; Mean Ratio Survival Time = 81, 95% CI 1-sided [lower limit 77.0], Standard Error of Mean 2.0 — Estimate is the ratio of the mean platelet survival time of treatment over control

3. Secondary Outcome: in Vitro Characteristics of Whole Blood and Platelets Derived From Mirasol-treated Whole Blood - Hemoglobin
Time Frame: Day 0 post-collection, day 0 post-illumination, day 1 post-storage
Population: Modified Intent to Treat population (mITT) = all enrolled subjects who signed informed consent and have valid data (excluding Subjects V01 through V08 who had irreparably confounded data due to a calibration error of the radioactivity detection device).
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Mirasol-treated Whole Blood: 1 unit of WB tested at the time of collection, immediately following Mirasol treatment, and 24 hours after Mirasol treatment.
Arm/Group | Mirasol-treated Whole Blood
Number analyzed (Participants) | 14
g/dL
  Day 0 post-collection | 12.49 (0.762)
  Day 0 post-illumination | 11.69 (0.741)
  Day 1 post-storage | 11.73 (0.732)

4. Secondary Outcome: in Vitro Characteristics of Whole Blood and Platelets Derived From Mirasol-treated Whole Blood - Hematocrit
Time Frame: Day 0 post-collection, day 0 post-illumination, day 1 post-storage
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of total blood volume
Arm/Group | Mirasol
Number analyzed (Participants) | 14
Percentage of total blood volume
  Day 0 post-collection | 35.88 (1.945)
  Day 0 post-illumination | 33.37 (1.754)
  Day 1 post-storage | 34.49 (1.691)

5. Secondary Outcome: in Vitro Characteristics of Whole Blood and Platelets Derived From Mirasol-treated Whole Blood - White Blood Cells
Time Frame: Day 0 post-collection, day 0 post-illumination, day 1 post-storage
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cells * 10e9/L
Arm/Group | Mirasol
Number analyzed (Participants) | 14
cells * 10e9/L
  Day 0 post-collection | 4.49 (1.002)
  Day 0 post-illumination | 4.17 (0.980)
  Day 1 post-storage | 3.64 (0.804)

6. Secondary Outcome: in Vitro Characteristics of Whole Blood and Platelets Derived From Mirasol-treated Whole Blood - Platelets
Time Frame: Day 0 post-collection, day 0 post-illumination, day 1 post-storage
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cells * 10e9/L
Arm/Group | Mirasol
Number analyzed (Participants) | 14
cells * 10e9/L
  Day 0 post-collection | 151.77 (43.051)
  Day 0 post-illumination | 110.52 (26.686)
  Day 1 post-storage | 154.43 (34.807)

7. Secondary Outcome: in Vitro Characteristics of Whole Blood and Platelets Derived From Mirasol-treated Whole Blood - pH
Description: pH is a measure of the acidity or alkalinity of a solution, numerically equal to 7 for neutral solutions, increasing with increasing alkalinity and decreasing with increasing acidity. The pH scale commonly in use ranges from 0 to 14
Time Frame: Day 0 post-collection, day 0 post-illumination, day 1 post-storage
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mirasol
Number analyzed (Participants) | 14
units on a scale
  Day 0 post-collection | 7.017 (0.0261)
  Day 0 post-illumination | 7.027 (0.0220)
  Day 1 post-storage | 6.804 (0.0256)

8. Secondary Outcome: in Vitro Characteristics of Whole Blood and Platelets Derived From Mirasol-treated Whole Blood - CO2
Time Frame: Day 0 post-collection, day 0 post-illumination, day 1 post-storage
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Mirasol
Number analyzed (Participants) | 14
kPa
  Day 0 post-collection | 9.96 (1.335)
  Day 0 post-illumination | 8.78 (0.946)
  Day 1 post-storage | 13.05 (1.216)

9. Secondary Outcome: in Vitro Characteristics of Whole Blood and Platelets Derived From Mirasol-treated Whole Blood - pO2
Time Frame: Day 0 post-collection, day 0 post-illumination, day 1 post-storage
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Mirasol
Number analyzed (Participants) | 14
kPa
  Day 0 post-collection | 5.93 (1.521)
  Day 0 post-illumination | 6.20 (2.069)
  Day 1 post-storage | 4.68 (1.146)

10. Secondary Outcome: in Vitro Characteristics of Whole Blood and Platelets Derived From Mirasol-treated Whole Blood - Potassium
Time Frame: Day 0 post-collection, day 0 post-illumination, day 1 post-storage
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Mirasol
Number analyzed (Participants) | 14
mmol/L
  Day 0 post-collection | 3.11 (0.192)
  Day 0 post-illumination | 3.10 (0.141)
  Day 1 post-storage | 5.86 (0.401)

11. Secondary Outcome: in Vitro Characteristics of Whole Blood and Platelets Derived From Mirasol-treated Whole Blood - Glucose
Time Frame: Day 0 post-collection, day 0 post-illumination, day 1 post-storage
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Mirasol
Number analyzed (Participants) | 14
mmol/L
  Day 0 post-collection | 20.50 (1.778)
  Day 0 post-illumination | 18.79 (1.498)
  Day 1 post-storage | 15.12 (1.625)

12. Secondary Outcome: in Vitro Characteristics of Whole Blood and Platelets Derived From Mirasol-treated Whole Blood - Lactate
Time Frame: Day 0 post-collection, day 0 post-illumination, day 1 post-storage
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Mirasol
Number analyzed (Participants) | 14
mmol/L
  Day 0 post-collection | 2.01 (0.635)
  Day 0 post-illumination | 2.44 (0.549)
  Day 1 post-storage | 8.97 (0.811)

13. Secondary Outcome: in Vitro Characteristics of Whole Blood and Platelets Derived From Mirasol-treated Whole Blood - Hemolysis
Description: Hemolysis is the rupture or destruction of red blood cells (RBCs), which releases hemoglobin from inside the RBCs into the plasma (where it is called "free hemoglobin"). Hemolysis is measured as the percentage of free hemoglobin compared to the total hemoglobin in a blood sample.
Time Frame: Day 0 post-collection, day 0 post-illumination, day 1 post-storage
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of free hemoglobin
Arm/Group | Mirasol
Number analyzed (Participants) | 14
percentage of free hemoglobin
  Day 0 post-collection | 0.1 (0.11)
  Day 0 post-illumination | 0.1 (0.10)
  Day 1 post-storage | 0.2 (0.10)

14. Secondary Outcome: in Vitro Characteristics of Whole Blood and Platelets Derived From Mirasol-treated Whole Blood - Plasma Free Hemoglobin
Time Frame: Day 0 post-collection, day 0 post-illumination, day 1 post-storage
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Mirasol
Number analyzed (Participants) | 14
g/L
  Day 0 post-collection | 0.24 (0.241)
  Day 0 post-illumination | 0.22 (0.204)
  Day 1 post-storage | 0.30 (0.211)

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | Mirasol
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 10/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirasol (N=22)
Hematoma (Injury, poisoning and procedural complications) | 5 (5)
Anxiety (Psychiatric disorders) | 2 (2)
Cold/influenza (Infections and infestations) | 1 (1)
Collapsed vein during donation (Vascular disorders) | 1 (1)
Vasovagal syncope (Nervous system disorders) | 1 (1)
Hypertension (Blood and lymphatic system disorders) | 1 (1)
Blisters on both feet (Skin and subcutaneous tissue disorders) | 1 (1)
Fever (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less